CLINICAL TRIAL: NCT02007590
Title: Does High-frequency Airflow Oscillation, Delivered Using Aerosure, Increase Exercise Capacity in Severe Chronic Obstructive Pulmonary Disease?
Brief Title: Aerosure and Six Minute Walk Distance in Severe COPD
Acronym: ACCORD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Actegy Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 13.LO.1124
Record Dates: First submitted 2013-12-06; First posted 2013-12-11 (Estimated); Last update posted 2018-01-11 (Actual); Status verified 2018-01

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Aerosure 25 Hz (Experimental): All subjects receive an active device, sham device (disabled) and no device in a randomised sequence.
  Interventions: Device: Aerosure 25 Hz
- Aerosure sham (Sham Comparator): All subjects receive an active device, sham device (disabled) and no device in a randomised sequence.
  Interventions: Device: Aerosure Sham
- No device (No Intervention): All subjects receive an active device, sham device (disabled) and no device in a randomised sequence.

INTERVENTIONS:
Device: Aerosure 25 Hz — Active Aerosure device
  Arms: Aerosure 25 Hz
Device: Aerosure Sham — Device designed to appear identical to active device but with HFAO mechanism disabled
  Arms: Aerosure sham

SUMMARY:
To investigate whether high frequency airflow oscillation (HFAO), delivered using Aerosure, increases six minute walk distance (6MWD) and reduces exertional breathlessness in patients with severe chronic obstructive pulmonary disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

* Stable severe COPD (FEV1 < 50% predicted)
* Modified MRC dyspnoea score 2 or greater
* At least 10 pack year smoking history
* Able to mobilise independently

Exclusion Criteria:

* Contraindications to spirometry [1]
* Contraindications to clinical exercise testing [2]
* Contraindications to HFAO (see section A.6.3b))
* Resting SpO2>88% on air or on patient's usual oxygen prescription
* Systolic arterial blood pressure (ABP) >200mmHg, diastolic ABP >100 mmHg

  1. Cooper, B.G., An update on contraindications for lung function testing. Thorax, 2010.
  2. ATS/ACCP Statement on Cardiopulmonary Exercise Testing. Am. J. Respir. Crit. Care Med., 2003. 167(2): p. 211-277.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-02; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Six minute walk distance (6MWD) | up to 6 minutes

SECONDARY OUTCOMES:
end-6MWD Borg breathlessness | after 6 minute walk test
Arterial oxygen saturation (SpO2) | At start of 6 minute walk test and after every 1 minute

OTHER OUTCOMES:
Inspiratory capacity (IC) | At end of 6 minute walk test

CONTACTS AND LOCATIONS:
Overall Officials: John Moxham, MD, Principal Investigator — King's College Hospital NHS Trust
Locations (1):
- King's College Hospital, Bessemer Road, Denmark Hill, London, United Kingdom